CLINICAL TRIAL: NCT03758222
Title: A Clinical Study to Evaluate the Safety and Feasibility (Including First in Human) of the XFLO EXPANDER SYSTEM (EXPANDER-1)
Brief Title: Safety and Feasibility of the XFLO Expander System (Mercury)
Acronym: EXPANDER-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MedeonBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-CIP-1164; PN-7585,-7998 10-MSC-1082 (Other: Prodeon Medical, Inc.)
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Arm-1: Device implantation for 1 month (Experimental): Treatment group receives intervention with the XFLO Expander System implantation for 1 month, and then retrieved.
  Interventions: Device: XFLO Expander System
- Arm-2: Device implantation for 6 months (Experimental): Treatment group receives intervention with the XFLO Expander System implantation for 6 months, and then retrieved.
  Interventions: Device: XFLO Expander System
- Arm-3: Device implantation for 12 months (Experimental): Treatment group receives intervention with the XFLO Expander System implantation for 12 months, and then retrieved.
  Interventions: Device: XFLO Expander System

INTERVENTIONS:
Device: XFLO Expander System — Implantation and retrieval of the XFLO Expander System in the prostatic urethra to treat benign prostatic hyperplasia (BPH)
  Other Names: Mercury

SUMMARY:
To demonstrate the safety and feasibility of the Mercury Expander system and procedure to treat patients with lower urinary tract symptoms (LUTS) secondary to urinary outflow obstruction from benign prostatic hyperplasia.

DETAILED DESCRIPTION:
A prospective, non-randomized, two-arm, multi-center clinical trial designed to evaluate the safety and feasibility of the Mercury Expander system in patients with lower urinary tract symptoms (LUTS) secondary to urinary outflow obstruction from benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Age ≥ 50 years
* Prostate volume 30 - 80 cc by Abdominal Ultrasound (AUS) or Trans Rectal Ultrasound (TRUS)
* Prostatic urethra length of 2.0-6.0 cm, as measured from bladder neck to verumontanum, using cystoscopy (or prostate length from bladder neck to external sphincter of 2.0-8.0 cm during screening visit, using ultrasound).
* Medication history

  * Not on BPH related medication for the past 6 months.
  * If on BPH related medication:

    * On 5-alpha-reductase inhibitors (ARIs), the patient must be on the medication for at least 3 months with a stable voiding pattern
    * On alpha-blockers, the patient must be on the medication for at least 3 weeks with a stable voiding pattern
* Patients with symptomatic BPH and related lower urinary tract symptoms (LUTS):

  * With International Prostate Symptom Score (IPSS) > 13; Qmax < 12 mL/sec on a voided volume ≥125 mL; Post-void residual (PVR) < 250 mL; QoL score ≥ 3

Exclusion Criteria:

* Previous BPH procedure
* Median prostatic lobe or high bladder neck
* Urethral stricture, meatal stenosis, or bladder neck obstruction - either current, or recurrent requiring 2 or more dilatations
* Elevated Prostate Specific Antigen (PSA) ≥ 10 ng/mL unless negative biopsy within last 6 months, or a positive biopsy showing cancer
* Cystolithiasis within the prior 3 months
* History of neurogenic bladder or urinary retention with PVR >1000mL.
* Serum creatinine >1.8 mg/dl or upper-tract disease which compromises renal function
* Current or recent Urinary Tract Infection (UTI) or disease
* Known allergy to nickel
* Life expectancy of less than 24 months
* Known coagulopathies or subject on anticoagulants or antiplatelets other than aspirin ≤ 100 mg (unless antiplatelets are withheld minimum 3 days prior to procedure)
* Anticipated need for additional surgery or treatments for comorbidities during the study period.
* Current gross hematuria
* Other co-morbidities that could impact the study results
* Unable or unwilling to complete all required questionnaires and follow-up assessments
* Unable or unwilling to sign informed consent form
* Currently enrolled in any other investigational clinical research trial that has not completed the primary endpoint.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Benign prostatic hyperplasia (BPH) is a male disease
Enrollment: 45 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Freedom from Unanticipated adverse device effects (UADEs) | 1 month (Arm-1)
  Measure any device or procedure related adverse events
Freedom from Unanticipated adverse device effects (UADEs) | 6 months (Arm-2)
  Measure any device or procedure related adverse events

SECONDARY OUTCOMES:
Freedom from Unanticipated adverse device effects (UADEs) | 7 months (Arm-1)
  Measure any device or procedure related adverse events
Freedom from Unanticipated adverse device effects (UADEs) | 12 months (Arm-2)
  Measure any device or procedure related adverse events
Change in International Prostate Symptom Score (IPSS) | 1 month and 7 months (Arm-1)
  Measure improvement in lower urinary tract symptoms related to benign prostatic hyperplasia (BPH)
Change in International Prostate Symptom Score (IPSS) | 6 and 12 months (Arm-2)
  Measure improvement in lower urinary tract symptoms related to benign prostatic hyperplasia (BPH)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Woo, MD, Principal Investigator — Australian Clinical Trials Pty Ltd
Locations (5):
- Australian Clinical Trials Pty Ltd, Wahroonga, New South Wales, Australia
- Canada (2):
  - University Health Network, Toronto, Ontario
  - Brunswick Medical Center, Montreal
- National Center of Urology, Tbilisi, Georgia
- China Medical University Hospital, Taichung, Taiwan